CLINICAL TRIAL: NCT00000208
Title: Methadone/Buprenorphine Cross-Over Study
Brief Title: Methadone/Buprenorphine Cross-Over Study - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-06082-4; R18-06082-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1993-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to explore ways to cross patients over from methadone to buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Opiate dependence according to DSM-IV critera. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hynotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-02

PRIMARY OUTCOMES:
Drug use
Withdrawal symptoms
Opiate craving

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Derived] Schurr MS, Chen YT, Raue PJ, Arean PA, Alexopoulos GS, Renn BN. Relation Between Executive Function Test Performance and Treatment Outcomes During Brief Psychotherapies for Later-Life Depression. Am J Geriatr Psychiatry Open Sci Educ Pract. 2025 Sep;7:1-11. doi: 10.1016/j.osep.2025.04.002. Epub 2025 Jun 11. PMID 41306470